CLINICAL TRIAL: NCT06853249
Title: Influence of Food Texture on Appetite Control, Gastric Emptying, and Energy Expenditure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anja Bosy-Westphal, Principal Investigator, Head of Department of Human Nutrition, University of Kiel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ABW-2025-YF
Record Dates: First submitted 2025-02-13; First posted 2025-02-28 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Nutrition; Healthy Male and Female Subjects
Keywords: food texture; appetite control; whole room indirect calorimetry (WRIC); energy balance; gastric emptying; ad libitum energy intake; liquid meals

STUDY DESIGN:
Intervention Model Description: The trial consists of two arms, each with two interventions. All participants will receive all interventions.
Who Masked: Participant
Masking Description: Blinding of participants to the actual primary outcome parameters to avoid energy intake bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- isocaloric preload (Experimental): In this arm of the study, participants receive two different isocaloric preloads for breakfast, one as a liquid meal and one as oatmeal.
  Interventions: Other: liquid meal; Other: semi-solid meal
- ad libitum preload (Experimental): In this arm of the study, participants are given two different isovolumetric drinks as a preload in addition to an ad libitum oatmeal breakfast. One drink is a liquid meal, the other is a non-caloric soft drink (water, sucralose, flavour).
  Interventions: Other: caloric drink + semi-solid meal; Other: non-caloric drink + semi-solid meal

INTERVENTIONS:
Other: liquid meal — An isocaloric amount (500 kcal) of a commercially available liquid meal with a matched macronutrient composition is consumed. After 5 hours, lunch is eaten ad libitum.
  Arms: isocaloric preload
Other: semi-solid meal — An isocaloric amount (500 kcal) of a commercially available semi-solid oatmeal with a matched macronutrient composition is consumed. After 5 hours, lunch is eaten ad libitum.
  Arms: isocaloric preload
Other: caloric drink + semi-solid meal — A predefined amount of a caloric drink (= liquid meal) together with an ad libitum amount of a semi-solid meal is consumed. After 5 hours, lunch is eaten ad libitum.
  Arms: ad libitum preload
Other: non-caloric drink + semi-solid meal — A predefined amount of a non-caloric drink (= water, sucralose, flavor) together with an ad libitum amount of a semi-solid meal is consumed. After 5 hours, lunch is eaten ad libitum.
  Arms: ad libitum preload

SUMMARY:
The aim of the study is to investigate the effect of liquid versus semi-solid meals on the regulation of energy balance in healthy young adults.The main questions it aims to answer are:

* Does a protein-rich liquid meal result in less satiety and therefore higher ad libitum energy intake at the next meal than an isocaloric oatmeal with the same macronutrient ratio?
* Is the consumption of a protein-rich liquid meal as a beverage in addition to an ad libitum oatmeal less compensated within the meal and at the next meal and provides thus a higher ad libitum energy intake than an isovolumetric noncaloric soft drink in addition to an ad libitum oatmeal?

Researchers will compare a protein-rich liquid meal to an isocaloric oatmeal with matched macronutrient composition to answer the first question. Researchers will compare a protein-rich liquid meal + oatmeal to a noncaloric softdrink (water with sucralose and flavoring) + oatmeal to answer the second question.

Participants will:

* spend 4 intervention days in a metabolic chamber (whole room indirect calorimeter)
* consume pre-definied preloads for breakfast and ad libitum lunch meals on 4 intervention days

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females
* Body Mass Index between 19-35 kg/m2
* low to medium habitual physical activity
* women with regular menstrual cycle (during intervention in follicular phase)

Exclusion Criteria:

* smoking (cigarettes + cannabis)
* chronic illnesses
* regular intake of medication
* Anemia and/or iron deficiency
* food allergies / intolerances
* vegans
* regular high physical activity (exercise >1 hour/d)
* current weight loss diet / weight loss of >5 kg in the last 3 months
* restraint eaters (according to the German version of the 'Three-Factor-Eating-Questionnaire', Stunkard und Messick (1985))
* active participation in another trial
* pregnant / lactating women
* persons incapable of giving informed legal consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female, male
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
ad libitum energy intake | for 9 hours after the consumption of the preloads
  measured during preload and lunch [kcal] following the preload in both arms

SECONDARY OUTCOMES:
gastric emptying | for 4 hours after the consumption of the isocaloric preloads
  gastric half-emptying time [min] determined with 13C-sodium acetate breath test, only assessed during arm "isocaloric preload"
eating rate at lunch | at 5 hours after consumption of the preload
  assessed during ad libitum lunch [g/min] following the preload in both arms
number of chews per bite at lunch | at 5 hours after consumption of the preload
  assessed during ad libitum lunch [number] following the preload in both arms
serum ghrelin concentrations | for 3 hours after consumption of the isocaloric preloads
  area under the serum ghrelin concentration curve over 3 hours
serum peptide-YY (PYY) concentrations | for 3 hours after consumption of the isocaloric preloads
  area under the serum PYY concentration curve over 3 hours
serum Glucagon-like Peptide 1 (GLP-1) concentrations | for 3 hours after consumption of the isocaloric preloads
  area under the serum GLP-1 concentration curve over 3 hours
energy expenditure | measured for 9.5 hours
  Measured as kcal for 9.5 hours in a whole room indirect calorimeter (WRIC), including the consumption of the preload and the ad libitum lunch.
macronutrient oxidation | measured for 9.5 hours
  Measured as respiratory exchange ratio (RER) for 9.5 hours in a whole room indirect calorimeter (WRIC), including the consumption of the preload and the ad libitum lunch.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, PhD, MD, Principal Investigator — University of Kiel, Department of Human Nutrition
Locations (1):
- Kiel University, Institute of Human Nutrition, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
Due to the privacy statement in the subject information form, data may not be publicly available but might be available upon reasonable request.